CLINICAL TRIAL: NCT04218578
Title: Association of Global Longitudinal Strain and Global Constructive Work With Cardiac Performance and Clinical Outcome One Year After MitraClip Implantation in Functional Mitral Regurgitation
Brief Title: Strain Imaging in Patients With Functional Mitral Regurgitation, Treated With MitraClip
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, associate professor, University of Athens
Other Study IDs: card,EBD308/10-05-2018
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Mitral Regurgitation; Heart Failure
Keywords: MitraClip; Functional mitral regurgitation; Reverse remodeling
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Device group: patients with heart failure and concomitant severe functional mitral regurgitation that were treated with MitraClip
  Interventions: Diagnostic Test: speckle tracking analysis of transthoracic echocardiogram
- Control group: patients with heart failure and concomitant severe functional mitral regurgitation that were treated with optimal medical treatment
  Interventions: Diagnostic Test: speckle tracking analysis of transthoracic echocardiogram

INTERVENTIONS:
Diagnostic Test: speckle tracking analysis of transthoracic echocardiogram — analysis at workstation with 2D strain-Speckle tracking echocardiography of transthoracic cardiac echo at baseline and one-year follow up examination

SUMMARY:
The aim of this study is i) to evaluate left ventricular global longitudinal strain and myocardial work in patients with heart failure and severe functional mitral regurgitation one year after MitraClip implantation and compare these variables with patients treated with optimal medical treatment and ii) to find echocardiographic predictors of clinical response and reverse left ventricular remodeling at one-year follow up.

DETAILED DESCRIPTION:
This study is one of the first in terms of publication. As far as the investigators know there are few papers with small series of patients regarding echocardiographic parameters and strain imaging in patients with functional mitral regurgitation (MR) and MitraClip. As the investigator's goal is to assess the potential impact of the MitraClip on myocardial deformation indexes, at the end of the study a direct comparison of changes of echocardiography markers -at one year follow up- between the control and device group will be performed. The changes in myocardial deformation markers will be associated with the respective changes in Brain-natriuretic peptide (BNP) levels, New York Heart Association (NYHA) class status, 6-minute walking distance (6MWD) and left ventricle (LV) volumes at follow -up. The investigators also aim to identify baseline prognostic echocardiography markers for the prediction of clinical improvement and LV reverse remodeling after successful edge-to-edge repair in functional MR patients during one year follow up. In specific, in this study the investigators will measure the 2-Dimension (2D) strain values of the left ventricle and left atrium (global longitudinal strain-GLS of the LV and Peak Atrial longitudinal strain - PALS of the left atrium) at baseline and at one year follow up, they will appreciate the LV myocardial work and all its components (Global Work Index-GWI, Global Constructed Work-GCW,Global wasted work-GWW and Global Work Efficiency-GWE) of the left ventricle and finally they will evaluate the baseline variables as predictors of reverse LV remodeling defined by reduction of left ventricle end-diastolic and end-systolic volume at one-year follow up.

ELIGIBILITY:
Inclusion Criteria:

* patients with EF more than 15% and below 45%
* Heart failure symptoms with NYHA class >2
* Moderate-to-severe and severe functional Mitral regurgitation

Exclusion Criteria:

* degenerative mitral regurgitation
* asymptomatic patients
* NYHA class IV patients not able to perform 6MWT
* EF>45%
* poor echocardiographic acoustic window patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart failure patients with severe functional mitral regurgitation that are treated either with MitraClip or with optimal medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Changes of LV volumes | one year
  change of left ventricular end-diastolic and end-systolic volumes during one-year follow up of the patients
Changes of NYHA class status | one year
  measurement of NYHA class status at baseline and one-year follow uo

SECONDARY OUTCOMES:
Changes of myocardial work of the LV | one year
  Evaluation of the components of myocardial work (Global work index, global constructive work, Global wasted Work and Global Work efficiency) at baseline and one-year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Professor, Study Chair — Attikon University Hospital of Athens
Locations (1):
- Attikon University Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Papadopoulos K, Ikonomidis I, Chrissoheris M, Chalapas A, Kourkoveli P, Parissis J, Spargias K. MitraClip and left ventricular reverse remodelling: a strain imaging study. ESC Heart Fail. 2020 Aug;7(4):1409-1418. doi: 10.1002/ehf2.12750. Epub 2020 May 20. PMID 32432839